CLINICAL TRIAL: NCT00163644
Title: Randomised Controlled Trial to Investigate the Effects of an Exercise Programme on Physical Performance and Quality of Life After a Bone Marrow Transplant
Brief Title: RCT to Investigate Whether an Exercise Programme Improves the Physical Performance and QOL After BMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: The Alfred (Other); The Leukaemia Foundation of Victoria (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 144/02
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Hematological Malignancies
Keywords: Hematological malignancies.; Bone- marrow/ haemopoetic transplant; Exercise
MeSH Terms: conditions — Hematologic Neoplasms; Motor Activity

ARMS (3):
- Aerobic exercise plus resistance (Active Comparator): Aerobic exercise plus resistance exercise for 6 weeks
  Interventions: Procedure: aereobic plus resisted exercise
- Aerobic exercise (Active Comparator): Aerobic exercise for 6 weeks
  Interventions: Procedure: aerobic plus active exercise
- Control (Other): No formal exercise and weekly phone calls
  Interventions: Other: No formal exercise plus phone calls

INTERVENTIONS:
Procedure: aereobic plus resisted exercise
  Arms: Aerobic exercise plus resistance
Procedure: aerobic plus active exercise
  Arms: Aerobic exercise
Other: No formal exercise plus phone calls
  Arms: Control

SUMMARY:
The hypothesis is that exercise will improve the physical performance and quality of life of bone marrow/ haemopoietic stem cell transplants.The aim of the trial is to provide definite clinical evidence as to which( if any) type of exercise is most beneficial for this patient population. It is also aimed at improving the provision of physiotherapy services to this group of patients.

DETAILED DESCRIPTION:
A three group, single blinded, randomised trial was designed to compare the effects of

1. aerobic plus active exercise and
2. aerobic plus resistance exercise to
3. control group of bone marrow/haemopoietic recipients not recieving exercise.

The hypotheses being tested is that

1. Exercise improves the physical performance of transplants recipients.
2. Exercise improves the quality of life of these patients;
3. resisted exercise added to aerobic exercise increases muscle strength or lean muscle mass and
4. There are no adverse events during either form of exercise

ELIGIBILITY:
Inclusion Criteria:

Recipient bone marrow transplant Alfred Hospital, Platelets >= 20 x 10E9 / l Provide written consent, 30 days after a bone marrow transplant have an absolute neutrophil count of 1x10E9/l be in a stable medical condition

Exclusion Criteria:

febrile neutropenia Have active graft versus host disease Have cardiomyopathy (ejection fraction < 20%) require > 28% oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2003-11; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Physical performance. | At 6 weeks
Quality of Life. | At 6 weeks
Anthropometry and Grip strength | At 6 weeks

SECONDARY OUTCOMES:
Heart Rate. | At 6 weeks
No adverse events during treatment. | At 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M Walsh, dip. physio, Principal Investigator — Bayside Health
Locations (1):
- Alfred hospital Physiotherapy dept,, Melbourne, Victoria, Australia